CLINICAL TRIAL: NCT05377749
Title: Families Addressing Cancer Together (FACT): A Pilot Randomized Trial
Brief Title: The Families Addressing Cancer Together Intervention for Parents With Cancer
Acronym: FACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LCCC2150; 5K07CA218167 (NIH)
Record Dates: First submitted 2022-04-20; First posted 2022-05-17 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Cancer; Parenting; Communication; Parents; Parent-Child Relations
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACT intervention (Experimental): Families Addressing Cancer Together (FACT) intervention plus questionnaires
  Interventions: Behavioral: FACT
- Wait-list control condition (No Intervention): Participants assigned to the waitlist control condition only complete questionnaires during the study period. After they have completed their 6-week study activities, they will receive access to the FACT intervention.

INTERVENTIONS:
Behavioral: FACT — Families Addressing Cancer Together (FACT) is a web-based intervention that provides tailored communication support for parents with cancer.
  Arms: FACT intervention

SUMMARY:
The proposed pilot randomized controlled trial will test the FACT (Families Addressing Cancer Together) intervention designed to improve parents' confidence and ability to talk about their cancer with their minor children. We will enroll 40 patients with cancer who have a minor child to participate in this single site, 6-week study. The primary hypothesis being tested is that an intervention that assists parents with their communication needs with their children can be feasible and acceptable when compared with a wait-list control condition.

DETAILED DESCRIPTION:
Parents with cancer are encouraged to be "honest and open" with their minor children about their illness. However, many lack access to professional support for their communication needs. Without this support, parents with cancer and their children experience avoidable psychosocial distress. In order to better support parental communication needs in cancer, psychosocial interventions that can be implemented across clinical practice settings are needed. To address this gap, we developed and pilot-tested FACT (Families Addressing Cancer Together) - a theory-guided, web-based psycho-educational intervention to help parents with cancer talk about their illness with their children in a developmentally appropriate way.

The proposed pilot randomized controlled trial will test the feasibility and acceptability of the FACT intervention. We will enroll 40 patients with cancer who have a minor child to participate in this single site, 6-week study. The primary hypothesis being tested is that an intervention that assists parents with their communication needs with their children can be feasible and acceptable when compared with a wait-list control condition. We will also explore preliminary effects of the intervention on parental communication and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent reviewed and signed;
* Age equal to or above 18 years;
* Ability to understand and comply with study procedures;
* Able to complete all study measures and visits in English;
* Be a parent (defined as biological, adoptive, foster, or step-parent), kin caregiver (defined as a relative or someone with a significant emotional relationship who provides full-time care and nurturing of a child), or legal guardian of a child age 3 to 17 years of age who can speak and understand English;
* Have a diagnosis of Stage II-IV (or equivalent) invasive solid tumor not in surveillance or survivorship

Exclusion Criteria:

* Unable to complete self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes;
* Prior participation in the pilot trial or development and user testing protocol preliminary to this study;
* No current or expected contact with their child; or
* Existence of other co-morbid disease, which in the opinion of the investigator, prohibits participation in the protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev M Nakamura, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 07/05/2022 through 02/22/2023 at one cancer center in North Carolina.
Pre-assignment Details: During this period, there have been 93 potential subjects who could be approached for screening. In total 47 subjects were found eligible for the study and started.
Groups:
- Families Addressing Cancer Together (FACT) Intervention: Families Addressing Cancer Together (FACT) intervention plus questionnaires
  FACT: Families Addressing Cancer Together (FACT) is a web-based intervention that provides tailored communication support for parents with cancer.
Period: Baseline Assessments
Arm/Group | Families Addressing Cancer Together (FACT) Intervention | Wait-list Control Condition
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0
Period: 3 Weeks
Arm/Group | Families Addressing Cancer Together (FACT) Intervention | Wait-list Control Condition
Started | 24 | 23
Completed | 21 | 18
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FACT Intervention | Wait-list Control Condition | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 15 | 15 | 30
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Families Addressing Cancer Together (FACT) Satisfaction Scale
Description: Acceptability was measured by the FACT satisfaction scale in the intervention group using the study-specific, 6-item FACT satisfaction scale. The total score range is 0-18 with higher scores indicating more satisfaction.
Time Frame: 3 weeks
Population: Participants who started the intervention and completed the post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Families Addressing Cancer Together (FACT) Intervention
Number analyzed (Participants) | 20
score on a scale | 16.24 (2.48)

2. Primary Outcome: Acceptability as Measured by FACT Satisfaction Scale
Description: Satisfaction with FACT will be measured in the intervention group using the study-specific, 6-item FACT satisfaction scale. Total score range is 0-18 with higher scores indicating more satisfaction.
Time Frame: 6 weeks
Population: Subjects joined to the study and completed satisfaction survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Families Addressing Cancer Together (FACT) Intervention: Families Addressing Cancer Together (FACT) intervention plus questionnaires.
  FACT: Families Addressing Cancer Together (FACT) is a web-based intervention that provides tailored communication support for parents with cancer.
Arm/Group | Families Addressing Cancer Together (FACT) Intervention
Number analyzed (Participants) | 23
score on a scale | 13.15 (1.83)

3. Primary Outcome: Acceptability as Assessed by a Semi-structured, Post-intervention Interview
Description: Satisfaction with FACT will be assessed via semi-structured, post-intervention interviews.
  Regarding n's, these interviews were offered as an optional part of participation among those randomized to the intervention (FACT). 12 participants agreed to participate in the interviews.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Positive: Reported positive overall experience.
- Beneficial: Described specific beneficial components
- Recommended: Recommended changes or suggestions
- Shortcomings: Identified shortcomings
Arm/Group | Positive | Beneficial | Recommended | Shortcomings
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Yes | 11 | 11 | 7 | 4
  No | 0 | 0 | 5 | 8
  Not reported | 1 | 1 | 0 | 0

4. Secondary Outcome: Recruitment Feasibility as Measured by Rate of Eligible Patients Who Consent to Study Participation
Description: Percentage of approached patients who meet study eligibility criteria who enroll (provide informed consent) in the study.
Time Frame: 6 weeks
Population: All participants were invited to the study including both arms.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Approaced: All participants were invited to the study including both arms.
Arm/Group | All Subjects Approaced
Number analyzed (Participants) | 93
Participants
  Number of Eligible Participants for Screening | 93
  Number of Participants Consented and Started | 47

5. Secondary Outcome: Feasibility of Participant Retention as Measured by Percentage of Participants Who Complete Survey
Description: Feasibility of participant retention as measured by the percentage of participants who complete at least one study survey, at the 3-week time point.
Time Frame: 3 weeks
Population: Participants who started the study and completed the post-intervention survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Families Addressing Cancer Together (FACT) Intervention | Wait-list Control Condition
Number analyzed (Participants) | 23 | 23
Participants | 21 | 18

6. Secondary Outcome: Feasibility of Participant Retention as Measured by Percentage of Participants Who Complete Survey Assessments at 6 Weeks.
Description: Percentage of enrolled participants who complete at least one study survey (any) at the 6-week time point.The number of participants who completed the assessment,
Time Frame: 6 weeks
Population: Subjects joined to the study and completed the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | FACT Intervention | Wait-list Control Condition
Number analyzed (Participants) | 24 | 23
Participants | 23 | 17

7. Secondary Outcome: Change From Baseline Communication Self-efficacy Using the CSES
Description: Change in parental communication self-efficacy will be measured using an adapted version of the Communication Self-Efficacy Scale (CSES). The 9-item CSES measures parental communication self-efficacy on a visual analogue scale, with a total score range of 0 to 100, with higher scores meaning more self-efficacy.
Time Frame: Baseline, 3 weeks
Population: Participants who started the study and completed the post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Families Addressing Cancer Together (FACT) Intervention | Wait-list Control Condition
Number analyzed (Participants) | 21 | 18
score on a scale | 6.46 (14.40) | 2.85 (9.28)

8. Secondary Outcome: Change From Baseline Communication Self-efficacy Using the CSES
Description: as for outcome 7
Time Frame: Baseline, 6 weeks
Population: Subjects who joined to the study and completed the assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACT Intervention | Wait-list Control Condition
Number analyzed (Participants) | 23 | 17
score on a scale | 9.47 (16.08) | 0.96 (14.10)

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment.
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
Arm/Group | FACT Intervention | Wait-list Control Condition
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT05377749/Prot_SAP_000.pdf